CLINICAL TRIAL: NCT02185391
Title: Development of Sustainable Methods in Interactive Patient Education to Improve Adherence After Cardiac Rehabilitation
Brief Title: Interactive Education of Patients With Coronary Heart Disease
Acronym: INSERT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Paracelsus Harz Clinic Bad Suderode. (Other)
Collaborators: The German Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: ParacelsusHCBS 2013-125
Record Dates: First submitted 2014-06-23; First posted 2014-07-09 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2015-04

CONDITIONS: Coronary Disease
Keywords: Coronary Disease; Audience Response System
MeSH Terms: conditions — Coronary Disease | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fact-finding group (Experimental): Intervention: Audience Response System and motivational telephone interview
  Interventions: Procedure: Audience Response System; Behavioral: Telephone interview
- control group (No Intervention)

INTERVENTIONS:
Procedure: Audience Response System — patients use during oral presentations an audience response system
  Arms: fact-finding group
Behavioral: Telephone interview — patients receive motivational telephone interviews after their residence in rehabilitation clinics
  Arms: fact-finding group

SUMMARY:
Coronary Heart Diseases are responsible for a high number of deaths in Germany. To determine the risk factors secondary prevention is of great importance. After their residence in rehabilitation centers patients often get rid of newly required skills. In addition to that parameters like BMI, blood pressure and cholesterol level return to their initial value.

Using an Audience Response System (ARS) during oral presentations in rehabilitation centers should improve the learning effect of patients. Furthermore patients will receive motivating telephone calls in the follow-up. These methods should lead to a sustainable improvement of learning effects, health care behavior and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Cardiovascular disease

Exclusion Criteria:

* Inability or refusal to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2014-05; Primary Completion 2014-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Training content as a measure of success | 3 - 4 weeks
  Reaching a total score (70 points) with respect to the training content as a measure of success of the current interactive patient education

SECONDARY OUTCOMES:
BMI and / or abdominal circumference | 12 months
  Change in BMI and / or abdominal circumference
Blood Cholesterol Values | 12 months
  Change in Blood Cholesterol Values
Depression Score | 12 months
  Change in Depression Score
Health Related Quality of Living | 12 months
  Change in Health Related Quality of Living
Stroke | 12 months
  Number of patients with a stroke
Myocardial Infarction | 12 months
  Number of patients with Myocardial Infarction

CONTACTS AND LOCATIONS:
Locations (1):
- Paracelsus Harz Clinic Bad Suderode, Quedlinburg, Saxony-Anhalt, Germany